CLINICAL TRIAL: NCT05283759
Title: UZ Brussel Heart Rhythm Management Center Monocentric Registry of Brugada Syndrome
Brief Title: UZ Brussel HRMC Registry of Brugada Syndrome
Acronym: HRMCBrS
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, Director of Heart Rhythm Management Center, Universitair Ziekenhuis Brussel
Other Study IDs: UZ Brussel Brugada registry
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood sample for DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention because it is a patient registry

SUMMARY:
The monocentric UZB registry for Brugada registry is intended to collect all data on patients affected by Brugada syndrome at UZ Brussel hospital (UZB).

DETAILED DESCRIPTION:
The monocentric UZB registry for Brugada registry is intended to collect all data on patients affected by Brugada syndrome.

These includes:

1. demographical data: age, sex
2. antropometric data: height, weight, BMI
3. clinical data: comorbidities, arrhythmias, PM or ICD implantation, therapy

3) data on the families: number of family members, sudden death history. 4) data on the genetics 5) data on: ECG, echocardiography, CT scan, MRI of heart, MRI of brain, ECG imaging, 3D electroanatomical mapping and ablation

ELIGIBILITY:
Inclusion Criteria:

* Brugada syndrome diagnosis

Exclusion Criteria:

* Other diagnosis different from Brugada syndrome

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brugada syndrome patients diagnosed following current guidelines: (Priori SG, Blomstrom-Lundqvist C, Mazzanti A, et al. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death the Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC) Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J 2015;36:2793-2867.) Both Brugada spontaneous type 1 and ajmaline induced will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1992-01-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias | through study completion, an average of 10 year
  Composite of: sudden cardiac death, aborted sudden cardiac death, ventricular fibrillation, sustained ventricular tachycardia, ICD appropriate therapy
Atrial fibrillation | through study completion, an average of 10 year
  Atrial fibrillation occurrence
Death for any cause | through study completion, an average of 10 year
  Death for any cause
Cardiovascular death | through study completion, an average of 10 year
  Death for cardiovascular cause
Genetic mutations | Baseline
  Genetic mutations (pathogenic and variant of unknown significance) associated with Brugada syndrome. Wide gene panel with next generation sequencing will be used: Roche SeqCap® EZ Human Exome Probes v3.0 for BrS.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel Heart Rhythm Management Center, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD sharing